CLINICAL TRIAL: NCT00815932
Title: The Effect of Transcranial Direct Current Stimulation (t-DCS) On the P300 Component of Event-Related Potentials in Patients With Chronic Neuropathic Pain Due To Complex Regional Pain Syndrome (CRPS) or Diabetic Neuropathy-A PILOT, DOUBLE-BLIND, SHAM-CONTROLLED, CROSS-OVER STUDY
Brief Title: The Effect of Transcranial Direct Current Stimulation (t-DCS) On the P300 Component of Event-Related Potentials in Patients With Chronic Neuropathic Pain Due To CRPS or Diabetic Neuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to unfixable problem in the research machine we had to withdrawn from the study
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Pesach Shvartzman, Head Department of Family Medicine, Soroka University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOR477808CTIL
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Diabetic Neuropathies; Complex Regional Pain Syndrome Type II; Resistant Peripheral Neuropathic Pain; Chemotherapy Induced Pain Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Causalgia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1-CRPS (Experimental): 10 tDCS naïve patients with CRPS-related neuropathic pain in upper limb
  Interventions: Device: TDCS/sham procedure on five consecutive days
- 2-DN (Experimental): 20 tDCS naïve patients with diabetic neuropathy
  Interventions: Device: TDCS/sham procedure on five consecutive days
- 3-RPNP (Experimental): 20 tDCS naïve patients with resistant peripheral neuropathic pain
  Interventions: Device: TDCS/sham procedure on five consecutive days
- 4-CIPN (Experimental): 10 tDCS naïve patients with CIPN-Chemotherapy Induced Pain Neuropathy patients
  Interventions: Device: TDCS/sham procedure on five consecutive days

INTERVENTIONS:
Device: TDCS/sham procedure on five consecutive days — The latency and amplitude of P300, subjective pain intensity, and pain thresholds for tactile and thermal stimuli will be determined at before and 15 min and 120 min after the 1st and 5th tDCS/sham procedure, To receive tDCS/sham treatment, two electrodes will be placed on the patient´s skull (for details see section Methods) and the patient will rest for 5 min. After that, the patient will receive 20 minutes of 2 mA tDCS/sham. Subjective pain intensity, and pain thresholds for tactile and thermal stimuli will be determined before-, 15 min after and 120 min after each tDCS/Sham procedure. At the 1st and 5th tDCS/Sham session, the latency and amplitude of P300 will be determined before-, 15 min after and 120 min after the tDCS/sham procedure.

SUMMARY:
This is a controlled trial designed to determine short- and long-term effects of repeated tDCS on the P300 component of event-related evoked potentials in patients with chronic neuropathic pain due to Complex regional Pain Syndrome (CRPS) or diabetic neuropathy as compared with healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* An affected upper limb or lower limb
* Diagnosed as : Diabetic neuropathy, Complex Regional Pain Syndrome (CRPS), Chemotherapy Induced Pain Neuropathy (CIPN), Peripheral Neuropathy.
* Have not responded to at least two medications of the following groups: Opioids. Tricyclics, SSRI, SNRI, Pregabalin, Gabapentin, Anticonvulsants.
* Positive LANSS or CRPS criteria as follows:

  1. Continuing pain which is disproportionate to any inciting event or for CRPS diagnosis.
  2. Must report at least one symptom (symptoms here are reports by subject) in each of the four following categories: sensory, vasomotor, sudomotor/edema, motor/trophic.
  3. Must display at least one sign (signs here refer to objective observation/testing) in in each of the four following categories: sensory, vasomotor, sudomotor/edema, motor/trophic;
* Must meet resistant neuropathic pain criteria - pain that is neuropathic in characters that at least two neuropathic medications not from the same group have been tried for at least a month without improvement or severe side-effects were experienced. Resistant neuropathic pain with a score for "average pain in the last 24 hours" ≥4 on a numeric scale 0-10
* tDCS naive

Exclusion Criteria:

* Serious health problems other than CRPS or resistant neuropathic pain (e.g. uncontrolled hypertension, uncontrolled diabetes, heart failure)
* Pain/painful conditions unrelated to CRPS or neuropathic pain
* Pregnancy
* History of seizures/epilepsy
* Implanted device (e.g. pacemaker)
* Active illicit drug/alcohol abuse
* Unable to follow directions or complete tools in Hebrew
* Previous exposure to tDCS stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Changes in the amplitude of P300 | 15 min after and 120 min after the 1st tDCS, 15 min after and 120 min after the 5st tDCS, and at the follow up 1 week after the 5th tDCS.
Changes in the Latency of P300 | 15 min after and 120 min after the 1st tDCS, 15 min after and 120 min after the 5st tDCS, and at the follow up 1 week after the 5th tDCS.

SECONDARY OUTCOMES:
Changes in Pain Intensity-will be calculated as the difference in scores on the 11-point numerical pain rating scale (0-10) | 15 min after and 120 min after each tDCS stimulation
Changes in Pain Thresholds for Tactile and Thermal Stimuli will be calculated as the difference between ratings obtained form pain threshold measurements before- and after tDCS | 15 min after and 120 min after each tDCS stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Pain and palliative care unit, Ben Gurion University of the Negev, Beersheba, Israel